CLINICAL TRIAL: NCT02512614
Title: Evaluation of Novel Antimicrobial Hand Towels
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCEZID-6102
Record Dates: First submitted 2015-06-24; First posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Diarrheal Diseases; Acute Respiratory Infections; Fever; Skin Infection
MeSH Terms: conditions — Fever; Cellulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparison (No Intervention): Hand hygiene education.
- Intervention (Experimental): Hand hygiene education and 4 antimicrobial hand towels
  Interventions: Other: Antimicrobial Hand Towel

INTERVENTIONS:
Other: Antimicrobial Hand Towel — Novel antimicrobial hand towel.
  Arms: Intervention

SUMMARY:
In March 2012, the investigators initiated a prospective, cluster-randomized, controlled field trial in Kisumu County, located in an area in western Kenya which has the highest under-five mortality rate in Kenya with 149 childhood deaths per 1,000 live births 9. The study was designed to evaluate the effectiveness of an antimicrobial hand towel (hereafter referred to as towel) in preventing diarrheal diseases, acute respiratory infections, self-reported fever, and skin infections in children <2 years old.

DETAILED DESCRIPTION:
In March 2012, the investigators initiated a prospective, cluster-randomized, controlled field trial in Kisumu County, located in an area in western Kenya which has the highest under-five mortality rate in Kenya with 149 childhood deaths per 1,000 live births 9. The study was designed to evaluate the effectiveness of an antimicrobial hand towel (hereafter referred to as towel) in preventing diarrheal diseases, acute respiratory infections (ARIs), self-reported fever, and skin infections in children <2 years old.

ELIGIBILITY:
Inclusion Criteria:

* Mother of a child <2 years old

Exclusion Criteria:

* Inaccessible enumeration area in the rainy season
* Multiple eligible children in a single compound
* Moved between census and round 1

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with diarrheal disease | Within 48 hours of enrollment
  The number of participants that experience 3 or more loose or watery stools

SECONDARY OUTCOMES:
Number of participants with respiratory infections | Within 48 hours of enrollment
Number of participants with a subjective fever | Within 48 hours of enrollment
Number of participants with a skin infection | Within 48 hours of enrollment